CLINICAL TRIAL: NCT02053974
Title: Protective Effects of Spironolactone Against Anthracycline Induced Cardiomyopathy
Brief Title: Spironolactone Against Anthracycline-induced Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Mahmut Akpek, Medical doctor of Cardiology department, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Makpek-1
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Anthracycline Induced Cardiotoxicity
Keywords: Anthracycline; spironolactone; cardiotoxicity
MeSH Terms: conditions — Cardiotoxicity | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spironolactone (Active Comparator): patients who randomized to spironolactone administered arm
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Patients who randomized to placebo administered arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Spironolactone — Spironolactone
  Other Names: 25 mg spironolactone orally
  Arms: Spironolactone
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study sought to investigate the whether spironolactone protects the heart against anthracycline-induced cardiotoxicity.

DETAILED DESCRIPTION:
Anthracyclines are the cornerstone in the treatment of numerous hematological and solid cancers. The most common side effect of anthracycline is cardiotoxicity and this may limits its use and increases the rate of mortality and morbidity. Cardiotoxicity is cumulative, dose dependent, and irreversible. Improvements in protective mechanisms against the cardiotoxicity of anthracycline are important to prevent the discontinuance of these chemotherapeutics.

Spironolactone is an aldosterone antagonist which blocks the last step of the rennin angiotensin aldosterone system (RAAS). The RAAS is one of the most effective systems in remodeling of the myocardium in post-myocardial damage. According to the RALES study, in patients with severe heart failure, 25 mg spironolactone per day in addition to the standard therapy has positive effects, particularly on cardiac fibrosis and on remodeling, and substantially reduces the risk of both morbidity and death. In the EPHESUS study, it has been shown that, after the myocardial damage due to infarction, the administration of aldosterone antagonists had positive effects on the remodeling process, left ventricular ejection fraction and primer end-points. In the present study, we tested the hypothesis that RAAS blockage with spironolactone may reduce the cardiotoxicity of anthracycline group chemotherapeutics.

ELIGIBILITY:
Inclusion Criteria:

* LVEF >50%
* first diagnosed breast cancer
* female sex

Exclusion Criteria:

* Prior breast cancer and/or prior anthracycline exposure history
* LVEF <50%
* Use of angiotensin converting enzyme inhibitors, angiotensin receptor blockers and beta blockers
* Creatinin value >2 mg/dl
* Presence of chronic kidney failure
* Potassium value >5.3 mg/dl
* Presence of adrenal gland diseases,
* Presence of severe liver failure
* Co-morbidities such as coronary heart disease, hypertension, atrial fibrillation, and valvular heart disease.
* Male patients were excluded for the homogenization of the study

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Decrease in left ventricular ejection fraction | 24 weeks on average

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Akpek, M.D., Principal Investigator — Erciyes University School of Medicine
Locations (1):
- Erciyes University School of Medicine, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Akpek M, Ozdogru I, Sahin O, Inanc M, Dogan A, Yazici C, Berk V, Karaca H, Kalay N, Oguzhan A, Ergin A. Protective effects of spironolactone against anthracycline-induced cardiomyopathy. Eur J Heart Fail. 2015 Jan;17(1):81-9. doi: 10.1002/ejhf.196. Epub 2014 Nov 20. PMID 25410653